CLINICAL TRIAL: NCT06648785
Title: Modified Capecitabine and Oxaliplatin (mCAPOX) for Patients With GI Malignancies
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Randall F Holcombe, Director-Faculty, University of Vermont Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003100/UVMCC2404
Record Dates: First submitted 2024-10-14; First posted 2024-10-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: GI Cancers
Keywords: capecitabine; oxaliplatin; GI; chemotherapy; fluoropyrimidine; modified schedule
MeSH Terms: interventions — Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Single arm pilot/feasibility design with tolerability and toxicity as primary endpoints and response as exploratory endpoint. Standard drug dosages utilized with no dose finding component to this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Modified administration schedule of capecitabine with oxaliplatin (Experimental): * Oxaliplatin (85mg/m2), will be administered IV every 2 weeks
  * Capecitabine (1000mg/m2) will be given twice daily, administered orally (PO) for 7 days, followed by 7 days with no capecitabine Cycles will repeat every 14 days.
  Interventions: Drug: oxaliplatin; Drug: Fluoropyrimidine

INTERVENTIONS:
Drug: oxaliplatin — 85 mg/m2 oxaliplatin
Drug: Fluoropyrimidine — oral fluoropyrimidine 1000mg/m2

SUMMARY:
This study is a single arm, non-randomized feasibility study with tolerability and toxicity evaluation as primary endpoints which seeks to determine if a modified administration schedule of capecitabine with oxaliplatin will result in less toxicity than standard FOLFOX or CAPOX regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patient with GI malignancy
* Provider plans non-curative intent treatment with either CAPOX or FOLFOX (mFOLFOX6) at standard dosages for >3 months NOTE: Patient is not required to have radiologically measurable disease. NOTE: Planned administration of other anti-cancer medications (eg bevacizumab, epidermal growth factor receptor antibodies, immunotherapy, tyrosine kinase inhibitors) is allowed.

Exclusion Criteria:

* Patients not meeting standard hematologic parameters for chemotherapy administration as follows:

  * Absolute neutrophil count (ANC) ≥ 1500
  * Platelet count ≥ 100,000 Patients not meeting standard liver function parameters for chemotherapy administration as follows:
  * AST ≤ 5x ULN
  * ALT ≤ 5X ULN
  * Total Bilirubin ≤ 1.5X ULN Patients not meeting standard renal function parameters for chemotherapy administration as follows:
  * Serum Creatinine ≤ 1.2 or creatinine clearance ≥ 30 ml/min NOTE: Planned administration of another cytotoxic chemotherapy (eg irinotecan) is an exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Tolerability | 115 days
  Number of toxicity-related treatment delays Number of dose reductions
Toxicity | 115 days
  Severity of acute oxaliplatin reactions, graded 1-4
Neuropathy | 2-4 months after therapy
  Neuropathy will be graded 1-4 after 2 &4 months of severity
Cytopenias | 115 days
  Frequency of cytopenia grade 3 or higher.

SECONDARY OUTCOMES:
Tumor response | 115 days
  Response rate after 3-4 months, with exact time of restaging per investigator choice and investigator usual practice

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No
Anonymized patient related data will be incorporated into publications and will be made available to other investigators at reasonable request.